CLINICAL TRIAL: NCT00462878
Title: MERONEM: Observational Study About Efficacy of Meropenem in Comparison of Meropenem and Glycopeptide in Treatment of Neutropenia Febrile in Allogenic Blood Stem Cell Transplantation Patients
Brief Title: Meropenem Versus Meropenem Plus Glycopeptide in Patients With Febrile Neutropenia After Allogenic Blood Stem Cell Transplantation
Acronym: MERONEM
Status: Completed | Type: Observational
Sponsor: PETHEMA Foundation (Other)
Responsible Party: Pethema, Pethema
Other Study IDs: 03-2002-GTA
Record Dates: First submitted 2007-04-18; First posted 2007-04-19 (Estimated); Last update posted 2009-05-12 (Estimated); Status verified 2009-05

CONDITIONS: Allogenic Blood Stem Cell Transplantation; Febrile Neutropenia
Keywords: Febrile neutropenia
MeSH Terms: conditions — Febrile Neutropenia | interventions — Meropenem; Vancomycin; Teicoplanin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Meropenem — antibiotic
Drug: Vancomycin — Antibiotic
Drug: Teicoplanin — Antibiotic

SUMMARY:
Observational study to compare the treatment in neutropenic patients after allogenic blood stem cell transplantation, with meropenem or meropenem plus glycopeptide.

DETAILED DESCRIPTION:
Observational study cost-effectivity to compare the treatment in neutropenic patients after allogenic blood stem cell transplantation, with meropenem or meropenem plus glycopeptide.

The study will be done in two consecutive cohorts of patients. First cohort: meropenem 1g/8h ev Second cohort: meropenem 1g/8h and glycopeptide (vancomycin 1g/12 h or teicoplanin 400 mg/24h)

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Patients submitted to allogenic transplant
* Neutropenia: neutrophils account < 500/mm3 or neutrophils account < 1000/mm3 with prevision to decrease until 500/mm3 at the next 24-48 h
* Signs and symptoms to infection
* Fever: Temperature> 38,3 ºC registered one time, or 38 ºC en two times separated 60 minutes in a period of 12 h.

Exclusion Criteria:

* Medical history of meropenem or glycopeptides hypersensitivity
* Renal failure or creatinine in serum > 2,25 mg/dl or creatinine clearance < 40 ml
* Liver insufficiency
* Childbearing potential or breast feeding period
* Contraindications to meropenem, vancomycin or teicoplanin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients submitted to allogenic transplant with neutropenia (neutrophils account < 500/mm3 or neutrophils account < 1000/mm3 with prevision to decrease until 500/mm3 at the next 24-48 h); Signs and symptoms to infection; Fever (Temperature> 38,3 ºC registered one time, or 38 ºC en two times separated 60 minutes in a period of 12 h)
Sampling Method: Non-Probability Sample
Enrollment: 392 (Estimated)
Dates: Start 2002-11; Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanz Miguel Angel, Doctor, Principal Investigator — Hospital La Fe
Locations (64):
- Spain (64):
  - Hospital Son Dureta, Palma de Mallorca, Balearic Islands
  - Hospital U. Germans Trias i Pujol, Badalona, Barcelona
  - Hospital C. de Barcelona, Barcelona, Barcelona
  - Hospital del Mar, Barcelona, Barcelona
  - Hospital Durant y Reynals, Barcelona, Barcelona
  - Hospital Sant Pau, Barcelona, Barcelona
  - Hospital U. Vall D'Hebron, Barcelona, Barcelona
  - Hospital General de Manresa, Manresa, Barcelona
  - Hospital Niño Jesus, Sabadell, Barcelona
  - Hospital Mutua Tarrasa, Terrassa, Barcelona
  - Hospital Insular de Las Palmas, Las Palmas de Gran Canaria, Canary Islands
  - Hospital Materno-Infantil de Las Palmas, Las Palmas de Gran Canaria, Canary Islands
  - Hospital Ntra Sra del Pino/Sabinal, Las Palmas de Gran Canaria, Canary Islands
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife, Canary Islands
  - Hospital Aránzazu, Santander, Cantabria
  - Hospital U. Marques de Valdecilla, Santander, Cantabria
  - Hospital General de Castellón, Castellon, Castellón
  - Hospital Puerta del Mar, Cadiz, Cádiz
  - Hospital Doctor Josep Trueta, Girona, Girona
  - H. Xeral de Galicia, A Coruña, La Coruña
  - Hospital Juan Canalejo, A Coruña, La Coruña
  - Hospital Virgen Blanca, León, León
  - Hospital Principe de Asturias, Alcalá de Henares, Madrid
  - Hospital Severo Ochoa, Leganés, Madrid
  - Clínica Puerta de Hierro, Madrid, Madrid
  - Hospital 12 de Octubre, Madrid, Madrid
  - Hospital Gregorio Marañón, Madrid, Madrid
  - Hospital La Paz, Madrid, Madrid
  - Hospital La Princesa, Madrid, Madrid
  - Hospital Ramón y Cajal, Madrid, Madrid
  - Hospital General de Murcia, Murcia, Murcia
  - Hospital Reina Sofia, Murcia, Murcia
  - Hospital U. Virgen de la Arrixaca, Murcia, Murcia
  - H. Universitario Virgen de la Victoria, Málaga, Málaga
  - Hospital Carlos Haya, Málaga, Málaga
  - Hospital Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Vírgen del Rocío, Seville, Sevilla
  - Hospital de Tarragona "Joan XXIII", Tarragona, Tarragona
  - Hospital Verge de la Cinta, Tortosa, Tarragona
  - Hospital de Sagunto, Sagunto, Valencia
  - Hospital Arnao de Vilanova, Valencia, Valencia
  - Hospital Dr. Peset, Valencia, Valencia
  - Hospital General U. de Valencia, Valencia, Valencia
  - Hospital U. La Fe, Valencia, Valencia
  - Instituto Valenciano de Oncología, Valencia, Valencia
  - Hospital Luis Alcañiz de Xátiva, Xàtiva, Valencia
  - Hospital C. de Valladolid, Valladolid, Valladolid
  - Hospital do Meixoeiro, Vigo, Vigo
  - Hospital C.U. De Zaragoza, Zaragoza, Zaragoza
  - Miguel Servet, Zaragoza, Zaragoza
  - Hospital G. de Alicante, Alicante
  - Hospital de la Ribera, Alzira
  - Basurtuko Ospitalea, Basurto
  - Hospital de Cruces, Bilbao
  - Hospital San Millan, Cáceres
  - Hospital Francesc de Borja, Gandia
  - Hospital Virgen de Las Nieves, Granada
  - Complexo H. Xeral-Calde, Lugo
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario Salamanca, Salamanca
  - Hospital Clínico Universitario de Santiago, Santiago de Compostela
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital U. La Fe (H. Infantil), Valencia
  - Hospital Rio Hortega, Valladolid

REFERENCES:
- [Background] Cometta A, Glauser MP. Empiric antibiotic monotherapy with carbapenems in febrile neutropenia: a review. J Chemother. 1996 Oct;8(5):375-81. doi: 10.1179/joc.1996.8.5.375. PMID 8957718
- [Background] Jarque I, Sanz MA. [Application of the concepts of evidence-based medicine to the evidence on the treatment of febrile neutropenia]. Enferm Infecc Microbiol Clin. 1999;17 Suppl 2:95-102. Spanish. PMID 10605194
- [Background] Klastersky J. Current attitudes for therapy of febrile neutropenia with consideration to cost-effectiveness. Curr Opin Oncol. 1998 Jul;10(4):284-90. doi: 10.1097/00001622-199807000-00002. PMID 9702394
- [Background] Hughes WT, Armstrong D, Bodey GP, Bow EJ, Brown AE, Calandra T, Feld R, Pizzo PA, Rolston KV, Shenep JL, Young LS. 2002 guidelines for the use of antimicrobial agents in neutropenic patients with cancer. Clin Infect Dis. 2002 Mar 15;34(6):730-51. doi: 10.1086/339215. Epub 2002 Feb 13. No abstract available. PMID 11850858
- [Background] Koya R, Andersen J, Fernandez H, Goodman M, Spector N, Smith R, Hanlon J, Cassileth PA. Analysis of the value of empiric vancomycin administration in febrile neutropenia occurring after autologous peripheral blood stem cell transplants. Bone Marrow Transplant. 1998 May;21(9):923-6. doi: 10.1038/sj.bmt.1701201. PMID 9613785
- [Background] Celebi H, Akan H, Akcaglayan E, Ustun C, Arat M. Febrile neutropenia in allogeneic and autologous peripheral blood stem cell transplantation and conventional chemotherapy for malignancies. Bone Marrow Transplant. 2000 Jul;26(2):211-4. doi: 10.1038/sj.bmt.1702503. PMID 10918433
- [Background] Smith TL, Pearson ML, Wilcox KR, Cruz C, Lancaster MV, Robinson-Dunn B, Tenover FC, Zervos MJ, Band JD, White E, Jarvis WR. Emergence of vancomycin resistance in Staphylococcus aureus. Glycopeptide-Intermediate Staphylococcus aureus Working Group. N Engl J Med. 1999 Feb 18;340(7):493-501. doi: 10.1056/NEJM199902183400701. PMID 10021469
- [Background] Dompeling EC, Donnelly JP, Deresinski SC, Feld R, Lane-Allman EF, De Pauw BE. Early identification of neutropenic patients at risk of grampositive bacteraemia and the impact of empirical administration of vancomycin. Eur J Cancer. 1996 Jul;32A(8):1332-9. doi: 10.1016/0959-8049(96)00050-0. PMID 8869095